CLINICAL TRIAL: NCT06095830
Title: Value of Blood Indices of Systemic Inflammation in Intensive Care Unit Patients With Abdominal Sepsis
Brief Title: Blood Indices of Systemic Inflammation in Critically Ill Patients With Abdominal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa AA Khaled, Prof., Assiut University
Other Study IDs: Abdominal sepsis in ICU
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Abdominal Sepsis; Critically Ill
Keywords: Blood indices of systemic inflammation
MeSH Terms: conditions — Intraabdominal Infections; Critical Illness | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients that recovered from sepsis without complications
  Interventions: Diagnostic Test: Complete blood count
- Group 2: Patients that didn't recover from sepsis.
  Further subdivided into:
  Group 2-A: developed complications Group 2-B: non-surviving
  Interventions: Diagnostic Test: Complete blood count
- Group 3: Control group of healthy individuals
  Interventions: Diagnostic Test: Complete blood count

INTERVENTIONS:
Diagnostic Test: Complete blood count — Complete blood count done on admission and on discharge for patients, from which the blood indices of systemic inflammation will be calculated and correlated with outcome

SUMMARY:
This study aims to clarify the role of blood indices of systemic inflammation in ICU-admitted patients with abdominal sepsis to assess their diagnostic significance as well as their prognostic value.

DETAILED DESCRIPTION:
Sepsis is a complex, multifactorial syndrome which can evolve into conditions of varying severity. If left untreated, it may lead to the functional impairment of one or more vital organs or systems. Severity of illness and the inherent mortality risk escalate from sepsis, through severe sepsis (defined as sepsis associated with at least one acute organ dysfunction, hypoperfusion, or hypotension) and septic shock up multi-organ failure. Previous studies have demonstrated that mortality rates increase dramatically in the event of severe sepsis and septic shock.

Abdominal infection is a common indication for admission to the intensive care unit (ICU) and the abdomen is the second most common site of invasive infection among critically ill patients in epidemiological and therapeutic studies. Abdominal infections are more often associated with septic shock and acute kidney injury than are infections in other sites. The spectrum of disease and severity is broad and management of these infections is challenging.

The inflammatory response in patients with sepsis depends on the causative pathogen and the host (genetic characteristics and coexisting illnesses), with differential responses at local, regional, and systemic levels.

On the systemic level, several indices have been used as a mirror to outcome in patients with various pathologies, of which are the Blood Indices of Systemic Inflammation.

As these blood indices are easy and available investigation that may be promising predictors in sepsis, we aim in this study to evaluate their role in abdominal sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 18 years old.
2. Patients fulfilling the Systemic Inflammatory Response Syndrome (SIRS) criteria.
3. Patients with an established diagnosis of abdominal sepsis, clinically and by investigations.

Exclusion Criteria:

1. Patients below the age of 18 years.
2. Patients with haematological disorders.
3. Patients with concomitant severe morbidity affecting the prognosis other than sepsis e.g. hypovolemic shock, brainstem infarction, pulmonary embolism, etc.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total sample size of 120 individuals
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of the prognostic value of blood indices of systemic inflammation | Baseline
  Correlate between the blood indices of systemic inflammation and the prognosis of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Abdelsattar, Prof, Study Director — Assiut University; Dina Hammad, Prof, Study Director — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt